CLINICAL TRIAL: NCT02111057
Title: Perioperative Flare in RA: Characterization of Clinical and Biological Features
Status: Completed | Type: Observational
Sponsor: Hospital for Special Surgery, New York (Other)
Responsible Party: Sponsor
Other Study IDs: 2014-233
Record Dates: First submitted 2014-04-08; First posted 2014-04-10 (Estimated); Last update posted 2019-10-21 (Actual); Status verified 2019-10

CONDITIONS: Rheumatoid Arthritis
Keywords: Rheumatoid Arthritis; Total Hip Replacement; Flare; Perioperative Outcomes
MeSH Terms: conditions — Arthritis, Rheumatoid

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — During surgery, the subjects' surgeon will take samples of the tissue removed as part of their surgery from their joint. Specifically for Total Hip Replacement (THR), the femoral head will be collected intraoperatively from standardized anatomic sites, (fovea and capsular reflection). For Total Knee replacement (TKR), tissue samples of the patella cartilage, distal femur and proximal tibia, and synovium from the suprapatellar pouch will be collected intraoperatively.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Perioperative RA: Patients with Rheumatoid Arthritis undergoing a primary or secondary total hip replacement, between the ages of 18 and 90.

SUMMARY:
Researchers at the Hospital for Special Surgery are trying to learn more about post-operative rheumatoid arthritis flare (RA). This study hopes to understand RA flare after total joint replacement surgery and what the result of flaring is for patients over the 6 weeks post operation.

Through this study we aim to describe rates, characteristics, and risk factors of RA flare within 6 weeks of total hip arthroplasty (THA) and total knee arthroplasty (TKA)

DETAILED DESCRIPTION:
The condition to be studied is worsening (flare) of rheumatoid arthritis (RA) in patients who have undergone arthroplasty. RA patients were recruited prior to elective THA and TKA and prospectively followed. Clinicians evaluated RA clinical characteristics 0-2 weeks before and 6 weeks post surgery. Patients answered questions regarding disease activity including self-reported joint counts and flare status weekly for 6 weeks.

ELIGIBILITY:
Inclusion Criteria:

1. Age >18
2. Patients with Rheumatoid Arthritis undergoing total joint replacement surgery
3. Satisfy American College of Rheumatology(ACR)/European League Against Rheumatism(EULAR) 2010 classification criteria and/or the 1987 RA criteria (see below) and be diagnosed with RA
4. For control subjects: Have OA(Osteoarthritis), SLE(Systemic lupus erythematosus) or other inflammatory arthritis.

Exclusion Criteria:

1. Diagnosis of any other systemic rheumatic disease
2. Diagnosis of or crystalline arthropathy.
3. Unable to understand or read English.
4. Unable to follow the study protocol in a reliable manner.
5. Age < 18 or >75.

EXPLANATION OF CRITERIA:

Rheumatoid arthritis 1987 criteria:

1. morning stiffness in and around joints lasting at least 1 hour before maximal improvement;
2. soft tissue swelling (arthritis) of 3 or more joint areas observed by a physician;
3. swelling (arthritis) of the proximal interphalangeal, metacarpophalangeal, or wrist joints;
4. symmetric swelling (arthritis);
5. rheumatoid nodules;
6. the presence of rheumatoid factor; and
7. radiographic erosions and/or periarticular osteopenia in hand and/or wrist joints.

   * Criteria 1 through 4 must have been present for at least 6 weeks. Rheumatoid arthritis is defined by the presence of 4 or more criteria, and no further qualifications (classic, definite, or probable) or list of exclusions are required.

ACR/EULAR 2010 criteria for the classification of RA:

Table 3. The 2010 American College of Rheumatology/European League Against Rheumatism classification criteria for rheumatoid arthritis

Target population (Who should be tested?): Patients who

1. have at least 1 joint with definite clinical synovitis (swelling)*
2. with the synovitis not better explained by another disease

Classification criteria for RA (score-based algorithm: add score of categories A-D;

a score of ≥6/10 is needed for classification of a patient as having definite RA

Score

A. Joint involvement

1 large joint 0

2-10 large joints 1

1-3 small joints (with or without involvement of large joints) 2

4-10 small joints (with or without involvement of large joints) 3

>10 joints (at least 1 small joint) 5

B. Serology (at least 1 test result is needed for classification)

Negative RF and negative ACPA 0

Low-positive RF or low-positive ACPA 2

High-positive RF or high-positive ACPA 3

C. Acute-phase reactants (at least 1 test result is needed for classification)

Normal CRP and normal ESR 0

Abnormal CRP or abnormal ESR 1

D. Duration of symptoms

< 6 weeks 0

* 6 weeks 1

  * The criteria are aimed at classification of newly presenting patients. In addition, patients with erosive disease typical of rheumatoid arthritis (RA) with a history compatible with prior fulfillment of the 2010 criteria should be classified as having RA. Patients with longstanding disease, including those whose disease is inactive (with or without treatment) who, based on retrospectively available data, have previously fulfilled the 2010 criteria should be classified as having RA.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population will comprise of roughly 200 patients with Rheumatoid Arthritis undergoing a total joint replacement.
Sampling Method: Non-Probability Sample
Enrollment: 162 (Actual)
Dates: Start 2013-10-16 (Actual); Primary Completion 2017-05-09 (Actual); Study Completion 2017-05-09 (Actual)

PRIMARY OUTCOMES:
Rate of RA Flare at 6 week post surgery | 6 weeks
  The primary outcome is the rate of RA flare within 6 weeks of surgery as measured by the Outcome Measures in Rheumatoid Arthritis Clinical Trials(OMERACT) flare questionnaire. For comparison, the rate of RA flare at 1 week post surgery is measured.

SECONDARY OUTCOMES:
Severity and impact of flares 6 weeks and one year post arthroplasty, using the OMERACT PFQs | 6 weeks and one year
  The OMERACT PFQs include flare intensity, duration of flare, worsening of domains associated with flare (pain, fatigue, stiffness, patient reported tender and swollen joint count, difficulties with coping and participation).

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital for Special Surgery, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Hospital for Special Surgery — http://www.hss.edu/
- See also: Principal Investigator, Susan Goodman MD — http://www.hss.edu/physicians_goodman-susan.asp

DOCUMENTS (2):
  • Informed Consent Form (2016-09-02): https://cdn.clinicaltrials.gov/large-docs/57/NCT02111057/ICF_000.pdf
  • Study Protocol and Statistical Analysis Plan (2017-03-09): https://cdn.clinicaltrials.gov/large-docs/57/NCT02111057/Prot_SAP_001.pdf